CLINICAL TRIAL: NCT06927453
Title: Assessment of the Effect of Covered Versus Uncovered Human Amniotic Membrane In Soft Tissue Healing During Alveolar Ridge Preservation: A Randomized Controlled Trial
Brief Title: Soft Tissue Healing During Alveolar Ridge Preservation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soft Tissue Healing
Record Dates: First submitted 2025-04-04; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-01

CONDITIONS: Badly Broken Maxillary Premolars Indicated for Extraction
Keywords: Human amniotic Membrane (HAM); Alveolar ridge preservation; Soft tissue healing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: blinding of outcome assessors and participants will be achieved as the different outcomes will be assessed for all groups by assessors other than the researchers doing the procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acrylic splint . (Active Comparator): ●The HAM particulate material will be packed into the extraction socket then the HAM will be tucked over the extraction socket then the socket plug will be maintained in place with approximating sutures using 5-0 resorbable suture material. The surgical site covered with the custom acrylic splint.
- No splint . (Active Comparator): The HAM particulate material will be packed into the extraction socket then the HAM will be tucked over the extraction socket then the socket plug will be maintained in place with approximating sutures using 5-0 resorbable suture material. The surgical site will not be covered by splint.

INTERVENTIONS:
Procedure: Acrylic splint — The HAM particulate material will be packed into the extraction socket then the HAM will be tucked over the extraction socket then the socket plug will be maintained in place with approximating sutures using 5-0 resorbable suture material. The surgical site covered with the custom acrylic splint.
Procedure: No splint — The HAM particulate material will be packed into the extraction socket then the HAM will be tucked over the extraction socket then the socket plug will be maintained in place with approximating sutures using 5-0 resorbable suture material. The surgical site will not be covered

SUMMARY:
Statement of the problem: Alveolar ridge preservation after tooth extractions is considered a challenge in oral surgery daily practice. Dental extraction is a traumatic procedure which leads to loss of alveolar bone. The alveolar bone remodeling, which occurs after tooth extraction, leads to vertical and horizontal bone volume loss. Although placentally derived allografts have been widely applied in medical procedures over the past 100 years, their use in the dental field is relatively new.

The aim of this study is to compare the effect of covering versus uncovering the HAM on soft tissue healing after alveolar ridge preservation procedure using customized splints.

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of covering versus uncovering the HAM on soft tissue healing after alveolar ridge preservation procedure using customized splints.

materials and methods: Careful extraction of the selected tooth will be performed. Then, the extraction sockets will be randomly allocated into two groups. The HAM particulate will be packed into the extraction socket as a standard method for both groups. Group A (n=24) socket will be covered with Human amnion membrane while group B (n=24) socket will be covered with the prefabricated acrylic splint. Soft tissue healing will be assessed (1ry outcome) every day for the first week, day after day second week, once in third and fourth week. Postoperative pain and swelling will be recorded daily by the patient for the 1st two weeks post surgically. Postoperative medication will be prescribed to the patient and postoperative instructions will be explained in detail. Follow-up will be performed to assess the parameters and to ensure performing proper oral hygiene. Data collected will be tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

1.Patients who need simple teeth extractions.

Exclusion Criteria:

1. Patients with inability or anticipated failure to maintain adequate oral hygiene.
2. Pregnant or breast-feeding mothers.
3. Any medical condition or therapy that can affect healing.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Soft tissue healing | every day for the first week, day after day second week, once in third and fourth week
  Surface area/intraoral Scanner in mm

SECONDARY OUTCOMES:
post operative pain | every day for the first week, day after day second week, once in third and fourth week
  Visual analog score ( score from 0 to 10 in which 0 is no pain and 10 is maximum pain )

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of oral and dental medicine , Suez university, Suez, Suez Governorate, Egypt